CLINICAL TRIAL: NCT04732754
Title: Effect of Cocoa Supplementation and Aerobic Exercise on Central Pressure and Arterial Stiffness Parameters in Physically Inactive Middle-aged Individuals
Brief Title: Effect of Cocoa Supplementation and Aerobic Exercise on Pressure Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP 5839.20
Record Dates: First submitted 2021-01-27; First posted 2021-02-01 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Sedentary Behavior
Keywords: Flavonoids; Cocoa; Arterial Stiffness; Physical Exercise; Central blood pressure
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Exercise; Control Groups; ASP protein, Theobroma cacao

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Double
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control Group (CG) (Placebo Comparator): This group will receive placebo capsules to be consumed for 8 weeks daily and will not exercise;
  Interventions: Dietary Supplement: Control Group (CG)
- Aerobic Exercise (AE) (Active Comparator): This group will receive placebo capsules and will perform 3 sessions of physical exercise / week, 50 min / session, with moderate intensity of 50-70% of VO2peak for 8 weeks.
  Interventions: Dietary Supplement: Aerobic Exercise (AE)
- Aerobic exercise + Theobroma cocoa (AETC) (Experimental): This group will receive 500mg cocoa capsules to be consumed daily and will perform 3 sessions of physical exercise / week, 50 min / session, with moderate intensity of 50-70% VO2peak) for 8 weeks
  Interventions: Dietary Supplement: Aerobic exercise + Theobroma cocoa (AETC)
- Theobroma cocoa (TC) (Experimental): This group will receive 500mg cocoa capsules to be consumed daily for 8 weeks.
  Interventions: Dietary Supplement: Theobroma Cocoa (TC)

INTERVENTIONS:
Dietary Supplement: Aerobic exercise + Theobroma cocoa (AETC) — Daily consumption of 500mg cocoa in capsules and 3 sessions of physical exercise / week, 50 min / session, with moderate intensity of 50-70% of VO2peak for 8 weeks.
  Arms: Aerobic exercise + Theobroma cocoa (AETC)
Dietary Supplement: Control Group (CG) — Daily consumption of placebo capsules for 8 weeks
  Arms: Control Group (CG)
Dietary Supplement: Aerobic Exercise (AE) — Daily consumption of placebo capsules and 3 sessions of physical exercise / week, 50 min / session, with moderate intensity of 50-70% of VO2peak for 8 weeks.
  Arms: Aerobic Exercise (AE)
Dietary Supplement: Theobroma Cocoa (TC) — Daily consumption of 500mg cocoa in capsules for 8 weeks.
  Arms: Theobroma cocoa (TC)

SUMMARY:
This study evaluates the cocoa supplementation and aerobic exercise on central pressure and arterial stiffness parameters in physically inactive middle-aged individuals.

500mg capsules will be offered to all patients. Of these, half will offer the content of 500mg of cocoa per capsule or placebo capsules. The placebo will contain a pharmacologically inert substance (microcrystalline cellulose) of the same color. A half will start 50' aerobic training 3 times/week while the other half will continue without exercise.

DETAILED DESCRIPTION:
Cardiovascular diseases (CVDs) are the number one cause of death in the world: more people die annually from CVDs than from any other cause. The arterial hypertension is one of the main predictors of CVDs. The number of adults with high blood pressure increased from 594 million in 1975 to 1.13 billion in 2015( WHO, 2020).

Due to the great increase in Hypertension around the world, new technological ways of assessing pressure have been discussed in the clinical setting, not only peripheral, but also central.

In this sense, the applanation tonometry of different arteries (carotid and radial), the analysis of pulses by various algorithms and the ability to estimate the shape of the pulse wave in the descending aorta root has been gaining prominence.

Flavonoids are a group of polyphenol compounds found in plants. The possible benefits from these compounds are related to cardiovascular health through specific actions on the artery wall. Prospective studies have shown that flavonoids can improve arterial stiffness, measured by Pulse Wave Velocity (PWV).

Physical exercise can intensifies organic functioning in different systems oh human body, including the cardiovascular. Studies has shown that chronic adaptations of pshysical exercise can improve arterial stiffness and central blood pressure parameters.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary lifestyle (IPAQ- International Physical Activity Questionnaire);
* Eutrophic or overweight (BMI >18,5kg/m² and <30kg/m²).

Exclusion Criteria:

* Individuals with a feverish state and / or infectious disease;
* Individuals with diabetes mellitus or coronary artery disease;
* Individuals who have any recent cardiovascular events (last 3 months) or chronic renal failure; history of malignant diseases with life expectancy <2 years;
* Use of statins;
* Smokers (those who have never smoked or smoked less than 100 cigarettes (5 bags of 20 cigarettes) in their lifetime and for at least 5 years);
* Alcoholics (The WHO estabilish ad acceptable the consumption is up to 15 doses / week for men and 10 for women, with 1 dose equivalent to approximately 350 mL of beer, 150 mL of wine or 40 mL of a distilled drink, considering that each contains between 10 and 15 g of ethanol);

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-12-10 (Estimated)

PRIMARY OUTCOMES:
Arterial Stiffness by Pulse Wave Velocity | 8 weeks
  The assessment of arterial stiffness will be carried out using the non-invasive method of PWV , which is obtained by dividing the carotid-femoral distance by the systolic wave travel time (in the unit of m / s) It will be checked by the Complior Analyzer equipment, with the volunteer in a supine position in an air-conditioned environment and controlled lighting in a LIC room, with the sensors placed over the right carotid and femoral arteries. The distance between the two points is measured by an infantometer and the data of pressure, total body weight and distance between the points of the sensors in the carotid artery and in the femoral artery are entered in the software to calculate the PWV. This analysis will be carried out before and after the intervention period.

CONTACTS AND LOCATIONS:
Overall Officials: Tainah Ortiz, M.Sc, Principal Investigator — Instituto de Cardiologia
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul/Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No